CLINICAL TRIAL: NCT00899847
Title: A Phase 2 Study of Autologous Followed by Nonmyeloablative Allogeneic Transplantation Using Total Lymphoid Irradiation (TLI) and Antithymocyte Globulin (ATG) in Multiple Myeloma Patients
Brief Title: Phase 2 Study of Autologous Followed by Nonmyeloablative Allogeneic Transplantation Using TLI & ATG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Wen-Kai Weng, Assistant Professor of Medicine (Blood and Marrow Transplantation), Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-15772; SU-04142009-2259 (Other: Stanford University); BMT201 (Other: OnCore Number)
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Results first posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-09

CONDITIONS: Transplantation, Homologous; Transplantation, Autologous; Multiple Myeloma; Blood and Marrow Transplant (BMT)
MeSH Terms: conditions — Multiple Myeloma | interventions — Transplantation; Filgrastim; Granulocyte Colony-Stimulating Factor; Cyclophosphamide; Melphalan; Cyclosporine; Antilymphocyte Serum; thymoglobulin; Mycophenolic Acid; Methylprednisolone Hemisuccinate; Calcium Dobesilate; Diphenhydramine; Acetaminophen; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | US Export: No

ARMS (1):
- Autologous-Allogeneic Peripheral Blood Stem Cell Transplant (Experimental): Study treatment is a high-dose sequential chemotherapy approach to hematopoietic stem cell (HSC) transplant that uses an autologous peripheral blood stem cell (auto-PBSC) transplant followed by allogeneic peripheral blood stem cell (allo-PBSC) transplant to evaluate improved graft vs host disease (GvHD) control. Participant auto-PBSC are mobilized with cyclophosphamide (also to provide cytoreduction) and filgrastim, followed by melphalan as an auto-PBSC conditioning agent, then auto-PBSC infusion. For the allo-PBSC transplant, donors are mobilized with filgrastim, and participants receive a regimen of total lymphoid irradiation and anti-thymocyte globulin (TLI/ATG), followed by infusion of donor allo-PBSC. Solumedrol, diphenhydramine, acetaminophen, and hydrocortisone are administered as premedications, and rabbit anti-thymocyte globulin (ATG) plus mycophenolate mofetil (MMF) are administered for post-allo-PBSC immunosuppression.
  Interventions: Procedure: Autologous peripheral blood stem cells (auto-PBSC) transplantation; Procedure: Allogeneic peripheral blood stem cells (allo-PBSC) transplantation; Drug: Filgrastim; Drug: Cyclophosphamide; Drug: Melphalan; Drug: Cyclosporine; Radiation: Total lymphoid irradiation; Biological: Rabbit anti-thymocyte globulin; Drug: Mycophenolate Mofetil 250mg; Drug: Solumedrol; Drug: Diphenhydramine; Drug: Acetaminophen; Drug: Hydrocortisone

INTERVENTIONS:
Procedure: Autologous peripheral blood stem cells (auto-PBSC) transplantation — Auto-PBSC ≥ 2 to 3 x 10e6 CD34+ cells/kg are intravenously (IV) infused as part of the combination stem cell therapy.
  and allogeneic stem cells are administered intravenous (IV) infusion to reestablish hematopoietic function in patients whose bone marrow or immune system is damaged or defective
  Other Names: auto-PBPC; Autologous peripheral blood progenitor cells (auto-PBPC) transplantation
Procedure: Allogeneic peripheral blood stem cells (allo-PBSC) transplantation — Allo-PBSC (target collection ≥ 5 x 10e6 CD34+ cells/kg) are intravenously (IV) infused as part of the combination stem cell therapy.
  Other Names: allo-PBSC; Allogeneic peripheral blood progenitor cells (allo-PBPC) transplantation
Drug: Filgrastim — Filgrastim is administered subcutaneously (SC) at 10 µg/kg/day for auto-PBSC mobilization starting day 2 of mobilization until the last day of apheresis.
  Filgrastim is administered SC at 5 µg/kg/day from Day 6 after auto-PBSC infusion to hematologic recovery.
  Filgrastim is administered SC at 16 µg/kg/day for donor allo-PBSC mobilization at from Day - 4 to Day 0, prior to allo-PBSC collection.
  Other Names: Neupogen; Granulocyte colony-stimulating factor (G-CSF); r-metHuG-CSF
Drug: Cyclophosphamide — Cyclophosphamide is administered intravenously (IV) at 4 g/m2 on Day 1 of the auto-PBSC mobilization regimen.
  Other Names: Ciclofosfamida; Ciclofosfamide; Claphene; CP monohydrate (CPM); CSP
Drug: Melphalan — Melphalan is administered after CSP at 200 mg/m2 intravenously (IV) on Day -2 before auto-PBSC infusion.
  Other Names: L-Sarcolysin; L-phenylalanine mustard (L-PAM); L-Sarcolysin phenylalanine mustard; L-sarcolysine
Drug: Cyclosporine — Cyclosporine is administered by mouth (PO) for allo-PBSC graft vs host disease (GvHD) prophylaxis at 5 mg/kg from Day -3 through Bay +56. Tacrolimus may substituted.
  Other Names: Cyclosporin; Cyclosporin A; Ciclosporin; CSP
Radiation: Total lymphoid irradiation — Total lymphoid irradiation is administered at 80 centigrey (cGy) on Day -11 to -7; and Day -4 to -2 before alllo-PBSC infusion. TLI is also administered at 80 centigrey (cGy) x 2 on Day -1 before alllo-PBSC infusion.
  Other Names: TLI
Biological: Rabbit anti-thymocyte globulin — ATG 1.5 mg/kg is administered intravenously (IV) on Day -11 to -7 before allo-PBSC infusion.
  Other Names: Thymoglobulin; ATG
Drug: Mycophenolate Mofetil 250mg — MMF is administered at 15 mg/kg 3x/day by mouth (PO) after allo-PBSC through Day 40, followed by 10% dose reduction weekly (dose taper) through day 96, and adjusted if there is evidence of MMF-related GI toxicity or excessive myelosuppression
  Other Names: CellCept; MMF
Drug: Solumedrol — Solumedrol 1 mg/kg is administered intravenously (IV) on Day -11 to -7 as a premedication for ATG and allo-PBSC infusion
  Other Names: Solumedin; Soludecadron
Drug: Diphenhydramine — Diphenhydramine 25 to 50 mg is administered as a premedication for the ATG; allo-PBSC; and DLI infusions.
  Other Names: Benadryl
Drug: Acetaminophen — Acetaminophen 650 mg is administered as a premedication for the ATG and allo-PBSC infusions.
  Other Names: Tylenol
Drug: Hydrocortisone — Hydrocortisone 100 mg is administered intravenously (IV) is a premedication for the allo-PBSC and DLI infusions.

SUMMARY:
To evaluate the toxicity and tolerability of this tandem autologous/allogeneic transplant approach for patients with advanced stage multiple myeloma.

DETAILED DESCRIPTION:
Development of cell-based immunotherapy from allogeneic hematopoietic cell transplantation (HCT) is dependent upon stable T-cell engraftment and the success of this therapeutic approach is likely to be greatest when directed against a minimal rather than gross tumor burden. To this end, tandem transplants with high dose therapy and autologous hematopoietic cell transplantation (AHCT) for tumor cytoreduction followed by non-myeloablative allotransplant have been conducted. In myeloma, this tandem approach results in greater efficacy compared to conventional AHCT.

ELIGIBILITY:
PARTICIPANT INCLUSION CRITERIA

* Stage II-III multiple myeloma or have progression after initial treatment of Stage I disease (Durie Salmon Staging). Patients with plasma cell leukemia are also included.
* Multiple myeloma / plasma cell leukemia diagnosis confirmed by pathology reviewed at Stanford University Medical Center.
* 18 to ≤ 75 years of age
* Karnofsky Performance Status > 70%.
* Corrected Carbon monoxide diffusing capacity (Dlco) > 60%
* Left ventricle ejection fraction (LVEF) > 50%.
* Alanine aminotransferase (ALT) ≤ 2 x normal
* Aspartate aminotransferase (AST) ≤ 2 x normal
* Total bilirubin ≤ 2 mg/dL, unless hemolysis or Gilbert's disease.
* Estimated creatinine clearance > 50 mL/min.
* Identified related or unrelated Human leukocyte antigen (HLA)-identical donor or donor with one antigen/allele mismatch in (HLA-A, B, C or DRB1).
* Signed informed consent.

DONOR INCLUSION CRITERIA

* At least 17 years of age
* HIV-seronegative
* Must be capable of giving signed, informed consent
* No contraindication to the administration of filgrastim
* Willing to have a central venous catheter placed for apheresis if peripheral veins are inadequate

PARTICIPANT EXCLUSION CRITERIA

* Prior allogeneic hematopoietic cell transplantation
* Uncontrolled active infection
* Uncontrolled congestive heart failure or angina
* HIV-positive
* Pregnant or nursing

DONOR EXCLUSION CRITERIA

* Serious medical or psychological illness
* Pregnant or lactating
* Prior malignancies within the last 5 years except for non-melanoma skin cancers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-05; Primary Completion 2014-04 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Kai Weng, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Autologous-Allogeneic Hematopoietic Stem Cell Transplant: Study treatment is a high-dose sequential chemotherapy approach to hematopoietic stem cell (HSC) transplant that uses an autologous peripheral blood stem cell (auto-PBSC) transplant followed by allogeneic peripheral blood stem cell (allo-PBSC) transplant to evaluate improved graft vs host disease (GvHD) control. Participant auto-PBSC are mobilized with cyclophosphamide (also to provide cytoreduction) and filgrastim, followed by melphalan as an auto-PBSC conditioning agent, then auto-PBSC infusion. For the allo-PBSC transplant, donors are mobilized with filgrastim, and participants receive a regimen of total lymphoid irradiation and anti-thymocyte globulin (TLI/ATG), followed by infusion of donor allo-PBSC. Solumedrol, diphenhydramine, acetaminophen, and hydrocortisone are administered as premedications, and rabbit anti-thymocyte globulin (ATG) plus mycophenolate mofetil (MMF) are administered for post-allo-PBSC immunosuppression.
Period: Overall Study
Arm/Group | Autologous-Allogeneic Hematopoietic Stem Cell Transplant
Started | 9
Completed | 7
Not Completed | 2
Not completed — Lack of suitable allogeneic donor | 2

BASELINE CHARACTERISTICS:
Groups:
- Autologous-Allogeneic Hematopoietic Stem Cell Transplant: A high-dose sequential chemotherapy approach with cyclophosphamide and etoposide followed by granulocyte colony stimulating factor (G-CSF) for collection of peripheral blood progenitor cells as well as for cytoreduction. Total Lymphoid irradiation and anti-thymocyte globulin (TLI/ATG).The preparatory regimens use BCNU and melphalan.
Arm/Group | Autologous-Allogeneic Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 54 [33 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Graft Versus Host Disease (GvHD)
Description: To evaluate the incidence acute GvHD of this tandem autologous/allogeneic transplant setting
Time Frame: 2 years after the last participant is enrolled.
Population: Due to the significance of the allo-PBSC transplant as a component to the treatment plan, participants who did not receive allo-PBSC are not included.
Measure: Count of Participants; unit: Participants
Arm/Group | Autologous-Allogeneic Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 7
Participants | 1

2. Secondary Outcome: Median Time to Engraftment After Auto-PBSC Transplant
Description: Engraftment is assessed as:
  * Neutrophil engraftment is > 0.5 x 10⁹/L after cytopenia
  * Platelet engraftment is > 20 x 10⁹/L after cytopenia
Time Frame: 1 month
Population: Includes all study participants
Measure: Median (Full Range); unit: Days
Arm/Group | Autologous-Allogeneic Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 9
Days
  Neutrophil Engraftment | 11 [10 to 12]
  Platelet Engraftment | 15 [10 to 20]

3. Secondary Outcome: Median Time to Engraftment After Allo-PBSC Transplant
Description: as for outcome 2
Time Frame: 1 month
Population: Due to the less intensive conditioning before allo-PBSC, only 2 participants experienced cytopenia, and thus only 2 participants could be evaluated for engraftment after allo-PBSC.
Measure: Median (Full Range); unit: Days
Arm/Group | Autologous-Allogeneic Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 2
Days
  Neutrophil Engraftment | 24 [24 to 24]
  Platelet Engraftment | 10 [10 to 10]

4. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall response rate (ORR) = Complete Response Rate (CRR) + Partial Response Rate (PRR)
Time Frame: 1 year
Population: Includes all study participants
Measure: Count of Participants; unit: Participants
Arm/Group | Autologous-Allogeneic Peripheral Blood Stem Cell Transplant
Number analyzed (Participants) | 9
Participants | 7

5. Secondary Outcome: Complete Response Rate (CRR)
Description: Complete response rate (CRR) was assessed as all of:
  * Negative immunoflixation on the serum and urine
  * Disappearance of any soft tissue plasmacytomas
  * < 5% plasma cells in bone marrow
Time Frame: 1 year
Population: Includes all study participants
Measure: Count of Participants; unit: Participants
Arm/Group | Autologous-Allogeneic Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 9
Participants | 3

6. Secondary Outcome: Partial Response Rate (PRR)
Description: Partial response rate (PRR) was assessed as
  * > 50% reduction in serum M-protein plus urine M-protein reduction by 90% or < 200 mg/24 hr
  * If serum M-protein is not measurable, then > 50% reduction in the involved serum free light chain
  * If involved serum free light chain is not measurable, then > 50% reduction in the bone marrow plasma cell percentage + > 50% reduction in the size of any soft tissue plasmacytoma.
Time Frame: 1 year
Population: Includes all study participants
Measure: Count of Participants; unit: Participants
Arm/Group | Autologous-Allogeneic Peripheral Blood Stem Cell Transplant
Number analyzed (Participants) | 9
Participants | 4

7. Secondary Outcome: Event-free Survival (EFS)
Description: To evaluate the graft versus myeloma effect by monitoring rate of event-free survival (EFS)
Time Frame: 2 years after the last participant is enrolled
Population: Includes all study participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Autologous-Allogeneic Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 9
percentage of participants | 44 [14 to 71]

8. Secondary Outcome: Overall Survival (OS)
Description: To evaluate the graft versus myeloma effect by monitoring rate of overall survival (OS)
Time Frame: 2 years after the last participant is enrolled
Population: Includes all study participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Autologous-Allogeneic Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 9
percentage of participants | 67 [28 to 87]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Autologous-Allogeneic Hematopoietic Stem Cell Transplant
Serious Adverse Events (participants affected / at risk) | 2/9
Other Adverse Events (participants affected / at risk) | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous-Allogeneic Hematopoietic Stem Cell Transplant (N=9)
Pulmonary Embolism (Vascular disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No